CLINICAL TRIAL: NCT02812654
Title: The Use of Ifosfamide, Doxorubicin and Hypofractionated Radiotherapy in Neoadjuvant Treatment of High-grade Extremity Soft Tissue and Non-metastatic Sarcomas
Brief Title: Ifosfamide, Doxorubicin and Hypofractionated Radiotherapy in Neoadjuvant Sarcoma Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1947/14
Record Dates: First submitted 2016-03-24; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-03

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma; soft tissue sarcoma; neoadjuvant chemotherapy; neoadjuvant radiotherapy; hypofractionated radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxorubicin, Ifosfamide, radiotherapy (Experimental): Doxorubicin 75mg/m2 (cycle 1,2 and 3), ifosfamide 9 g/m2 (cycle 1 and 3) and radiotherapy: 25 Gy / 5 x 500 cGy/day, beginning at Cycle2/Day1. The surgery will performed after 4-6 weeks from cycle 3. The remain viable cells in surgical specimen will be analyzed and if it accounts less than 30% the patient will receive more 3 cycles of cT. A boost of RT is indicated if margins are considered R1.
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide; Radiation: radiotherapy

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 75mg/m2 (cycle 1,2 and 3)
  Other Names: Adriamycin
Drug: Ifosfamide — Ifosfamide 9 g/m2 (cycle 1 and 3)
  Other Names: Mitoxana
Radiation: radiotherapy — radiotherapy: 25 Gy / 5 x 500 cGy/day

SUMMARY:
Prospective phase II study. Patients will be submitted to neoadjuvant chemotherapy (cT) and hypo fractionated radiotherapy (hRT) following by surgery. The remain viable cells will be analyzed and the patients whithin less than 30% will receive more 3 cycles of cT. All patients have deep high grade soft tissue sarcoma of extremity.

DETAILED DESCRIPTION:
Prospective phase II non controlled study. Staging: All patients will be submitted to a local Magnetic Resonance (MR), Chest Tomography (CT) and Positron emission tomography-computed tomography (PET CT) previous to treatment. After the first cT cycle a new PET CT will be provided and one more at the end of the neoadjuvant treatment. Chemotherapy: cT neoadjuvant: Doxorubicin 75mg/m2 (cycles 1,2 and 3), and ifosfamide 9 g/m2 (cycles 1 and 3). Radiotherapy: RT 25 Gy / 5 x 500 cGy/day, beginning at Cycle 2/Day1. The surgery will be performed after 4-6 weeks from cycle 3. The remain of viable cells in surgical specimen will be analyzed and whether the the percentage value is less than 30% the patient will receive more 3 cycles of cT. A boost of RT is indicated if margins are considered R1 (microscopic positive margin).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-75 years old, with non metastatic deeply high grade soft tissue sarcoma of extremities. KPS > 70% (Karnofsky Performance Status Score)

Exclusion Criteria:

* Patients with rhabdomyosarcoma, neuroendocrine tumor (Pnet) and chondrosarcomas, or who have had received radiotherapy (RT) or chemotherapy (cT) previous, or recurrent tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate disease free survival after neoadjuvant treatment | 24 months
  Evaluate local and distant disease free survival after the treatment

SECONDARY OUTCOMES:
Evaluate wound complication rates | 30 days
  Evaluate if this treatment is comparable with the Institution previous results using only cT as neoadjuvant treatment (20% of wound complications).
Amputation rates | 30 days
  Evaluate if it can be maintained the amputation rate (less than 5%)
cT morbidity | 6 months
  Evaluate the morbidity rates related to cT scheme

OTHER OUTCOMES:
PET CT response | 3 months
  Evaluate if the SUV (Standard uptake value) varies after first and third cycle and if it is related to survival

CONTACTS AND LOCATIONS:
Overall Officials: Ademar Lopes, Phd, Principal Investigator — A.C.Camargo Cancer Center
Locations (1):
- A.C.Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aguiar Junior S, Ferreira Fde O, Rossi BM, Santos EM, Salvajoli JV, Lopes A. Neoadjuvant chemoradiation therapy for soft tissue sarcomas of the extremities. Clinics (Sao Paulo). 2009;64(11):1059-64. doi: 10.1590/S1807-59322009001100005. PMID 19936179
- [Background] Aguiar S Jr, da Cunha IW, Lopes A. Genomic expression, chemotherapy response, and molecular targets in soft tissue sarcomas of the extremities: promising strategies for treatment selection. J Surg Oncol. 2010 Jan 1;101(1):92-6. doi: 10.1002/jso.21422. PMID 19834919
- [Background] Benz MR, Czernin J, Allen-Auerbach MS, Tap WD, Dry SM, Elashoff D, Chow K, Evilevitch V, Eckardt JJ, Phelps ME, Weber WA, Eilber FC. FDG-PET/CT imaging predicts histopathologic treatment responses after the initial cycle of neoadjuvant chemotherapy in high-grade soft-tissue sarcomas. Clin Cancer Res. 2009 Apr 15;15(8):2856-63. doi: 10.1158/1078-0432.CCR-08-2537. Epub 2009 Apr 7. PMID 19351756
- [Background] Cormier JN, Huang X, Xing Y, Thall PF, Wang X, Benjamin RS, Pollock RE, Antonescu CR, Maki RG, Brennan MF, Pisters PW. Cohort analysis of patients with localized, high-risk, extremity soft tissue sarcoma treated at two cancer centers: chemotherapy-associated outcomes. J Clin Oncol. 2004 Nov 15;22(22):4567-74. doi: 10.1200/JCO.2004.02.057. PMID 15542808
- [Background] Eilber FC, Rosen G, Nelson SD, Selch M, Dorey F, Eckardt J, Eilber FR. High-grade extremity soft tissue sarcomas: factors predictive of local recurrence and its effect on morbidity and mortality. Ann Surg. 2003 Feb;237(2):218-26. doi: 10.1097/01.SLA.0000048448.56448.70. PMID 12560780
- [Background] Freedman GM. Hypofractionated radiation therapy in the treatment of early-stage breast cancer. Curr Oncol Rep. 2012 Feb;14(1):12-9. doi: 10.1007/s11912-011-0207-7. PMID 22071682
- [Background] Grobmyer SR, Maki RG, Demetri GD, Mazumdar M, Riedel E, Brennan MF, Singer S. Neo-adjuvant chemotherapy for primary high-grade extremity soft tissue sarcoma. Ann Oncol. 2004 Nov;15(11):1667-72. doi: 10.1093/annonc/mdh431. PMID 15520069
- [Background] Gronchi A, Frustaci S, Mercuri M, Martin J, Lopez-Pousa A, Verderio P, Mariani L, Valagussa P, Miceli R, Stacchiotti S, Dei Tos AP, De Paoli A, Longhi A, Poveda A, Quagliuolo V, Comandone A, Casali PG, Picci P. Short, full-dose adjuvant chemotherapy in high-risk adult soft tissue sarcomas: a randomized clinical trial from the Italian Sarcoma Group and the Spanish Sarcoma Group. J Clin Oncol. 2012 Mar 10;30(8):850-6. doi: 10.1200/JCO.2011.37.7218. Epub 2012 Feb 6. PMID 22312103
- [Derived] Gobo Silva ML, Lopes de Mello CA, Aguiar Junior S, D'Almeida Costa F, Stevanato Filho PR, Santoro Bezerra T, Nakagawa SA, Nascimento AG, Werneck da Cunha I, Spencer Sobreira Batista RM, Nicolau Daher UR, Da Cruz Formiga MN, Germano JN, Catin Kupper BE, De Assis Pellizzon AC, Lopes A. Neoadjuvant hypofractionated radiotherapy and chemotherapy for extremity soft tissue sarcomas: Safety, feasibility, and early oncologic outcomes of a phase 2 trial. Radiother Oncol. 2021 Jun;159:161-167. doi: 10.1016/j.radonc.2021.03.033. Epub 2021 Mar 31. PMID 33798613
- [Derived] Spencer RM, Aguiar Junior S, Ferreira FO, Stevanato Filho PR, Kupper BE, Silva ML, Mello CA, Bezerra TS, Lopes A. Neoadjuvant Hypofractionated Radiotherapy and Chemotherapy in High-Grade Extremity Soft Tissue Sarcomas: Phase 2 Clinical Trial Protocol. JMIR Res Protoc. 2017 May 25;6(5):e97. doi: 10.2196/resprot.6806. PMID 28546135